CLINICAL TRIAL: NCT00290004
Title: Phase I/II Trial of Weekly Motexafin Gadolinium (MGd) for Patients With Refractory or Relapsed Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Study of Weekly Motexafin Gadolinium (MGd) for Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0223
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Leukemia; Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Leukemia; Lymphoma; Motexafin Gadolinium; Relapsed Chronic Lymphocytic Leukemia; Relapsed Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: motexafin gadolinium

SUMMARY:
The primary purpose of this study is to evaluate the safety, toxicities, dosage and response rate for an investigational drug, motexafin gadolinium, administered to patients with chronic lymphocytic leukemia or small lymphocytic lymphoma. The secondary purpose of this study is to evaluate the clinical benefit rate, the time it takes for a patient's chronic lymphocytic leukemia or small lymphocytic lymphoma to worsen, the duration of response and the time during which patients survive without chronic lymphocytic leukemia or small lymphocytic lymphoma worsening. Additionally, the patient's response to motexafin gadolinium will be compared to the response of the patient's cells in a laboratory to motexafin gadolinium.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* CLL as defined by the NCI 96 criteria (exception; patients may have bright surface immunoglobulin staining if negative for t[11;14] translocation or cyclin D1) or SLL as defined by WHO classification criteria and is refractory or relapsed as defined by one of the following:

  * Refractory disease: progressive disease while on therapy
  * Relapsed disease: progressive disease after at least one treatment course of therapy with disease response or stabilization
* ECOG performance status score of 0, 1, or 2
* Willing and able to provide written informed consent

Exclusion Criteria:

* Laboratory values of:

  * Platelet count < 30,000/µL
  * AST or ALT > 2 x ULN (upper limit of normal)
  * Total bilirubin > 2 x ULN
  * Creatinine > 2 mg/dL
* Chemotherapy, radiation therapy, immunotherapy, systemic corticosteroids (> 10 mg oral prednisone or equivalent), or systemic biologic anticancer therapy within 21 days before beginning study treatment
* Major surgery or hospitalization for a serious illness within the last 3 months
* Greater than three prior regimens (where a regimen is defined as a treatment for CLL/SLL given initially or after disease progression)
* Prior malignancy requiring current or prior treatment within the past 5 years, except for cervical neoplasia in situ and non-melanomatous skin cancer
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Phase I
To determine the maximum tolerated dose (MTD) of MGd when administered once weekly to patients with relapsed or refractory CLL/SLL
To determine the dose-limiting toxicities (DLTs) of MGd when administered once weekly to patients with relapsed or refractory CLL/SLL
Phase II
To assess the complete and partial response rate in patients with relapsed or refractory CLL/SLL when administered MGd once weekly at the MTD

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Evens, DO, Principal Investigator — Robert H. Lurie Comprehensive Cancer Center of Northwestern University; Neil E Kay, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - USC Norris Cancer Hospital, Los Angeles, California
  - Scripps Cancer Center, San Diego, California
  - Northwestern University, Chicago, Illinois
  - The Mayo Clinic, Rochester, Minnesota